CLINICAL TRIAL: NCT07310069
Title: A Phase II, Single-Arm, Multicenter Study of Gemcitabine and Nab-Paclitaxel in Combination With Iparomlimab and Tuvorilimab in Patients With Advanced Gallbladder Cancer
Brief Title: Gemcitabine and Nab-Paclitaxel Combined With Iparomlimab and Tuvorilimab for Advanced Gallbladder Cancer
Acronym: TRANSFORM-GBC
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Wei Gong, MD., Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XHEC-C-2025-111-4
Record Dates: First submitted 2025-12-01; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Gallbladder Cancer Unresectable
Keywords: gallbladder cancer
MeSH Terms: conditions — Gallbladder Neoplasms | interventions — 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Intervention Model Description: Gemcitabine plus Nab-Paclitaxel (AG regimen) in combination with Iparomlimab and Tuvorilimab (a dual anti-PD-1/CTLA-4 bispecific antibody)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment :Gemcitabine plus Nab-Paclitaxel (AG regimen) in combination with Iparomlimab and Tuvorili (Experimental): Treatment :Gemcitabine plus Nab-Paclitaxel (AG regimen) in combination with Iparomlimab and Tuvorili
  Interventions: Drug: Treatment :Gemcitabine plus Nab-Paclitaxel (AG regimen) in combination with Iparomlimab and Tuvorili

INTERVENTIONS:
Drug: Treatment :Gemcitabine plus Nab-Paclitaxel (AG regimen) in combination with Iparomlimab and Tuvorili — Treatment :Gemcitabine plus Nab-Paclitaxel (AG regimen) in combination with Iparomlimab and Tuvorili

SUMMARY:
This is a single-arm, multicenter, Phase II clinical trial evaluating the efficacy and safety of Gemcitabine plus Nab-Paclitaxel (AG regimen) in combination with Iparomlimab and Tuvorilimab (a dual anti-PD-1/CTLA-4 bispecific antibody) in patients with advanced unresectable gallbladder cancer.

The study aims to assess the surgical conversion rate and objective response rate (ORR) as primary endpoints. Secondary endpoints include R0 resection rate, disease control rate (DCR), progression-free survival (PFS), overall survival (OS), and safety profiles.

A total of 44 participants will be enrolled across three centers in China. The study is scheduled to run from May 2025 to April 2027.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Age 18-75 years.
* ECOG performance status 0-2, Child-Pugh class A.
* Histologically or cytologically confirmed advanced gallbladder cancer, deemed unresectable for R0 resection.
* Adequate organ function:
* ANC ≥1.5×10⁹/L, platelets ≥75×10⁹/L, hemoglobin ≥90 g/L.
* Serum creatinine ≤1.2 mg/dL or creatinine clearance ≥60 mL/min.
* Total bilirubin ≤1.5×ULN (≤3×ULN if liver metastases); AST/ALT ≤3×ULN (≤5×ULN if liver metastases).
* Life expectancy ≥3 months.
* Non-pregnant, non-lactating women and willingness to use contraception during and for 3 months after treatment.

Exclusion Criteria:

* Severe systemic infection or uncontrolled comorbidities (e.g., heart failure, thyroid disease, psychiatric disorders); active autoimmune disease requiring medication.
* Known allergy or intolerance to chemotherapy agents.
* Prior antitumor therapy (chemotherapy, radiotherapy, immunotherapy) within the past year, or history of other malignancies (except cured cervical carcinoma in situ or non-melanoma skin cancer).
* Pregnancy, lactation, or unwillingness to use contraception.
* Participation in another clinical trial within 30 days before the first dose.
* Unwillingness to participate or inability to provide informed consent.
* Any other condition that, in the investigator's judgment, may affect patient safety or compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
ORR | At the end of Cycle 6 (each cycle is 21 days)
  The objective response rate (ORR) of this quadruplet regimen as first-line therapy
Surgical Conversion Rate | At the end of Cycle 6 (each cycle is 21 days)
  Proportion of patients who achieve successful conversion to radical resection (R0/R1) after systemic therapy.

SECONDARY OUTCOMES:
Downstaging Rate | At the end of Cycle 6 (each cycle is 21 days)
  Proportion of patients whose clinical stage is reduced after conversion therapy.
Pathologic Response Rate | At the end of Cycle 6 (each cycle is 21 days)
  Proportion of patients with pathologic downstaging or major pathologic response in resected specimens
R0 Resection Rate | At the end of Cycle 6 (each cycle is 21 days)
  Proportion of patients who undergo R0 resection among those who receive surgery.
Disease Control Rate (DCR) | At the end of Cycle 6 (each cycle is 21 days)
  Proportion of patients with CR, PR, or stable disease (SD) lasting ≥4 weeks.
Recurrence-Free Survival (RFS) | up to 2 years
  Proportion of patients without recurrence at 2 years after resection.
Overall Survival (OS) | through study completion,up to 3 years
  Time from enrollment to death from any cause.
Adverse Events (AEs) / Serious AEs (SAEs) | through study completion, up to 30 days
  Incidence and severity of AEs and SAEs graded by CTCAE v5.0.
Surgical Safety | Perioperative
  Incidence of surgery-related complications (e.g., infection, bleeding, organ dysfunction)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Gong, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No